CLINICAL TRIAL: NCT05590039
Title: Prospective Clinical Study To Evaluate The Safety And Efficacy Of The MyEllevate® Procedure
Brief Title: Study To Evaluate The Safety And Efficacy Of The MyEllevate® Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7053-PL01-2022
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Soft Tissue Approximation; Elevation of Subdermis; Elevation of Underlying Muscle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment for MyEllevate Procedure (Experimental): The subjects were treated with the MyEllevate procedure.
  Interventions: Device: MyEllevate Procedure

INTERVENTIONS:
Device: MyEllevate Procedure — The defined study area will be identified and may be marked with a surgical marker.
  A local tumescent anesthetic, such as lidocaine, will be injected to the area prior to the procedure. The MyEllevate® device will be used in accordance with the Instructions for Use (IFU) manual for soft tissue approximation and elevation of sub dermis and underlying muscle of the submentum and jawline.

SUMMARY:
The intended purpose of the MyEllevate® procedure used in this study is to assess the safety and efficacy of the procedure for soft tissue approximation and elevation of sub dermis and underlying muscle of the submentum & jawline.

DETAILED DESCRIPTION:
Subjects are to be enrolled in this clinical study if they are a healthy male or female between the age of 18 - 65. Up to 10 subjects will be enrolled at 2 study centers. All subjects will attend a screening/pre-procedure visit which may be performed on the same day as the procedure visit but no more than 30 days prior to their procedure.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female between the age of 18 - 65.
* Must have any or all the following: visible platysma bands, glands and/or sagging in the submentum, jawline and/or neck.
* Reads and understands English.
* Understands and accepts obligation not to receive any other procedures on the treatment area through the length of the study.
* Understands and accepts the obligation and is logistically able to be present for all visits.
* Is willing to comply with all requirements of the study and sign the informed consent document.

Exclusion Criteria:

Is pregnant or of childbearing potential and not using medically effective birth control, or has been pregnant in the last 3 months, currently breast feeding or planning a pregnancy during the study.

* Is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within in the area to be treated 6 months (or at the discretion of the Investigator) prior to entering this study.
* Have received any treatments or procedures (including injectables such as Botox or fillers) in the area to be treated at least 4 months prior to treatment.
* Take antiplatelets, anticoagulants, thrombolytics, or anti-inflammatories.
* Have an active localized or systemic infection.
* Have an open wound in area being treated.
* Have a significant systemic illness or an illness localized in area being treated.
* Have had recent surgeries or problems in the treatment area (e.g. neck fracture, neck sprain, pinched nerve, spondylosis, arthritis in the neck).
* Have a history of thrombophlebitis.
* Have a history of heart failure or kidney disease.
* Have a history of allergic reaction or intolerance to the anesthesia used during the procedure.
* Have a history of poor wound healing.
* Have a history of poor circulation.
* Have a systemic autoimmune disease known to impair wound healing.
* Have a history of keloid formation.
* Currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within the area to be treated 6 months (or at the discretion of the Investigator) prior to entering this study.
* Has any condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound study results or may interfere significantly with the subject's participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Canavan, Study Director — Cynosure, Inc.
Locations (2):
- United States (2):
  - New Jersey Plastic Surgery, Montclair, New Jersey
  - Aesthetic Pavilion Ambulatory Surgery Center, Staten Island, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gupta V, Sharma VK. Skin typing: Fitzpatrick grading and others. Clin Dermatol. 2019 Sep-Oct;37(5):430-436. doi: 10.1016/j.clindermatol.2019.07.010. Epub 2019 Jul 17. PMID 31896400

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment for MyEllevate Procedure: The subjects were treated with the MyEllevate procedure.
  MyEllevate Procedure: The defined study area will be identified and may be marked with a surgical marker.
  A local tumescent anesthetic, such as lidocaine, will be injected to the area prior to the procedure. The MyEllevate® device will be used in accordance with the Instructions for Use (IFU) manual for soft tissue approximation and elevation of sub dermis and underlying muscle of the submentum and jawline.
Period: Overall Study
Arm/Group | Treatment for MyEllevate Procedure
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment for MyEllevate Procedure
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Fitzpatrick Skin Types [Count of Participants; unit: Participants] — Fitzpatrick Skin Types range from I-VI, with I meaning little melanin and light hair, and VI representing high amounts of melanin and dark hair. Additional details on this scale can be found in the publication cited for the results section.
  Participants
    Fitzpatrick Skin Type I | 1
    Fitzpatrick Skin Type II | 2
    Fitzpatrick Skin Type III | 5
    Fitzpatrick Skin Type IV | 2
    Fitzpatrick Skin Type V | 0
    Fitzpatrick Skin Type VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Physician Global Aesthetic Improvement Score (PGAIS)
Description: The physician will grade the improvement that they see at the 30 day follow up (30 days post treatment). They will grade them as one of the following: Very Much Improved, Much Improved, Improved, No Change, or Worsened.
Time Frame: 30 days post last treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment for MyEllevate Procedure
Number analyzed (Participants) | 10
Participants
  Very Much Improved | 5
  Much Improved | 3
  Improved | 2
  No Change | 0
  Worsened | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected until 90 days post treatment.
Arm/Group | Treatment for MyEllevate Procedure
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment for MyEllevate Procedure (N=10)
Bruising (Skin and subcutaneous tissue disorders) | 3
Edema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Pain/tenderness (Skin and subcutaneous tissue disorders) | 1
Skin discoloration (Skin and subcutaneous tissue disorders) | 1
Skin redundancy (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT05590039/Prot_SAP_000.pdf